CLINICAL TRIAL: NCT03523845
Title: Etiology of Early Apical Peri-implantitis: A Case-control Study Over a 20-year Period.
Brief Title: Etiology of Early Apical Peri-implantitis
Acronym: EAP
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Miguel Peñarrocha Diago, Head of Oral Surgery and Implantology. Medical and Dental School, Universitat of València, Spain., University of Valencia
Other Study IDs: LPI1
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Early Apical Peri-implantitis
Keywords: "early apical peri-implantitis"; "implant periapical lesion"; "retrograde peri-implantitis"; "implant failure"

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group: Test group (patients diagnosed with early apical peri-implantitis diagnosed)
  Interventions: Other: Observational intervention to diagnose an early apical peri-implantitis
- Control group: Control group (patients whose implants had not developed any inflammatory/infectious process and were osseointegrated)
  Interventions: Other: Observational intervention to diagnose an early apical peri-implantitis

INTERVENTIONS:
Other: Observational intervention to diagnose an early apical peri-implantitis — diagnose an early apical peri-implantitis

SUMMARY:
A case-control study was performed was performed following the STROBE statement from 1996 to 2016 including patients who were diagnosed with early apical peri-implantitis. Data were collected at the time of implant placement, and once the patients developed signs and symptoms consistent with early apical peri-implantitis, to determine the frequency and etiology of this pathology.

DETAILED DESCRIPTION:
A case-control study was performed following the STROBE statement (17) at the Oral Surgery Department, Faculty of Medicine and Dentistry (University of Valencia, Spain) from 1996 to 2016, in which patients with early peri-implantitis diagnosed were included (Figure 1). All patients were informed about the study design and procedures. Prior to participating, they were requested to sign an informed consent document. The study design was approved by the Ethical Committee of the University of Valencia (H1478255958653).

Two groups were established: Test group (patients diagnosed with early apical peri-implantitis diagnosed) and Control group (patients whose implants had not developed any inflammatory/infectious process and were osseointegrated).

ELIGIBILITY:
Inclusion Criteria:

* The following inclusion criteria were applied: patients ≥18 years old and controlled medical conditions who received treatment with implants. Additionally, for the test group, inclusion criteria were: symptoms and signs suggesting early apical peri-implantitis after implant placement; absence of implant mobility; dull percussion of nonsurmerged implants; presence or absence of radiolucency apically.

Exclusion Criteria:

* for the both groups: implants placed with guided bone regeneration or inadequate follow-up for failing to maintenance visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who received at least one dental implant
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 1996-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
type of surgery | Intraoperative
  immediate/delayed placement
tooth-implant distance | Intraoperative
  mesial and distal tooth-implant distance measured at the apex
Tooth status | Intraoperative
  apical lesion or endodontic treatment in the tooth being replaced or adjacent tooth endodontically treated

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Peñarrocha Diago, MD, MDM, PhD, Study Chair — Professor and Chairman of Oral Surgery and Implantology. Medical and Dental School, Universitat of València, Spain; Juan Antonio Blaya Tárraga, DDS, MSc, Principal Investigator — Master of Oral Surgery and Implantology

IPD SHARING:
Plan to Share IPD: Undecided
higher permissions are needed to make the decision

REFERENCES:
- [Background] Quirynen M, Gijbels F, Jacobs R. An infected jawbone site compromising successful osseointegration. Periodontol 2000. 2003;33:129-44. doi: 10.1046/j.0906-6713.2002.03311.x. No abstract available. PMID 12950847
- [Result] Lefever D, Van Assche N, Temmerman A, Teughels W, Quirynen M. Aetiology, microbiology and therapy of periapical lesions around oral implants: a retrospective analysis. J Clin Periodontol. 2013 Mar;40(3):296-302. doi: 10.1111/jcpe.12045. Epub 2012 Dec 27. PMID 23278599
- [Result] Penarrocha-Diago M, Maestre-Ferrin L, Cervera-Ballester J, Penarrocha-Oltra D. Implant periapical lesion: diagnosis and treatment. Med Oral Patol Oral Cir Bucal. 2012 Nov 1;17(6):e1023-7. doi: 10.4317/medoral.17996. PMID 22926472
- [Result] Zhao D, Wu Y, Xu C, Zhang F. Immediate dental implant placement into infected vs. non-infected sockets: a meta-analysis. Clin Oral Implants Res. 2016 Oct;27(10):1290-1296. doi: 10.1111/clr.12739. Epub 2015 Dec 15. PMID 26667097